CLINICAL TRIAL: NCT03674346
Title: Efficacy of Hypnoanalgesia by a Radiological Radiologist Technologist in Children With Cutaneous Angioma Treated With Sclerosis in Interventional Radiology
Brief Title: Efficacy of Hypnoanalgesia by a Radiologist Technologist in Children With Cutaneous Angioma Treated With Sclerosis in Interventional Radiology
Acronym: HYP-ANGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0044
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Angioma
Keywords: hypnoanalgesia; cutaneous angioma; sclerosis treatment
MeSH Terms: conditions — Hemangioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnoanalgesia group (Experimental): It is performed by a radiologist technologist who has been trained in Ericksonian hypnoanalgesia in the Hospices Civils de Lyon and has been practicing it regularly for 1 year.
  Interventions: Other: Hypnoanalgesia group
- MEOPA Group (Other): The pain management will be done exclusively by a mask delivering the equimolecular mixture of oxygen and nitrous oxide (MEOPA)
  Interventions: Other: Meopa Group

INTERVENTIONS:
Other: Hypnoanalgesia group — The running of a hypnosis session is protocolized and is based on three times:
  * The hypnotic induction time that allows to move from the state of consciousness to a modified state of consciousness: it will be adapted according to the patient as specified by the procedure of Ericksonian hypnosis. It varies from a few seconds to 10 minutes. Induction time depends on the patient's level of stress, apprehension, subsequent experiences of hospitalization, history, and level of hypnotizability.
  * The dissociation time. It is the state of modified consciousness obtained at the end of the induction which is prolonged,
  * The time of "return". It is time that allows the patient to regain his classic state of consciousness.
  Arms: Hypnoanalgesia group
Other: Meopa Group — The pain management will be done exclusively by a mask delivering the equimolecular mixture of oxygen and nitrous oxide (MEOPA) throughout the procedure.
  For optimal use, the beginning of its administration by the radiological technologist is performed 3 minutes before the sclerosant injection (at the end of the locating ultrasound). The end of administration will correspond to the end of the injections of the sclerosing product. These sclerosing products are not considered experimental or ancillary products in this study.
  Arms: MEOPA Group

SUMMARY:
This study highlights the global management of the various components of outpatient pain by hypnoanalgesia (pain management by hypnosis) in radiopediatrics.

Indeed, pain is induced by sclerosis of cutaneous angiomas in interventional radiology. It is managed by MEOPA (an equimolar mixture of oxygen nitrous oxide) or by general anesthesia.

For four years, the medical electroradiology technologist of the Mother and Child Hospital (HFME) of the Hospices Civils de Lyon offer patients in addition a pain management by hypnoanalgesia.

The investigator propose a multicenter open randomized study comparing two pain management strategies, in children aged 7 to 18 years treated for cutaneous angioma by sclerosis in interventional radiology at the HFME. The two strategies studied are: Hypnoanalgesia and MEOPA (the reference strategy).

The main objective is to evaluate the efficacy of hypnoanalgesia compared to the standard of care of pain, which is the use of MEOPA, in the treatment of sclerosis of cutaneous angioma in pediatric interventional radiology.

ELIGIBILITY:
Inclusion Criteria:

* Child requiring a first treatment with sclerosis cutaneous angioma whose location allows treatment in interventional radiology room,
* Child from 7 to 18 years old on the day of treatment,
* Free and informed consent of the child and his parents (or legal representative),
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Child under tutorship or guardianship,
* Child suffering from severe psychotic disorders or under psychotropic drug treatment,
* Child who has already had angioma sclerosis in the interventional radiology room. Indeed, the child can remember a previous support and have a priori, positive or negative, on the new support (memory bias),
* Child not speaking French,
* Deaf child or hearing impaired not allowing easy listening

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 138 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
assessment of pain score by Visual Analog Scale (EVA) | Day 0
  Comparison of the pain score felt by the child during the procedure (score 0 or 1, absence or presence of pain, on an Analog Visual Scale (EVA)) between the MEOPA group and the hypnoanalgesia group.

SECONDARY OUTCOMES:
Patient anxiety score assessed by anxiety Visual Analog Scale (EVA) | Day 0
number of side effects | Day 0
  comparaison between groups.
gravity of side effects | Day 0
  comparaison between groups.
Patient satisfaction assessed by a satisfaction questionary | Day 0
Pain assessed by Visual Analog Scale (EVA) | Day 0
anxiety assessed by Visual Analog Scale (EVA) | Day 0
number of injections performed per site | Day 0
MEOPA administration time | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Claire BENOIT-RUBY, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No